CLINICAL TRIAL: NCT01075776
Title: The Effects of C-type Natriuretic Peptide on Endothelial Function Following Ischaemia-Reperfusion in the Human Forearm
Brief Title: The Effects of C-type Natriuretic Peptide on Human Forearm Blood Vessels
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Queen Mary University of London (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Amrita Ahluwalia, Professor of Vascular Pharmacology, Queen Mary University of London
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 007143
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Ischaemia-reperfusion (IR) Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — Natriuretic Peptide, C-Type; Sodium Chloride; Acetylcholine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CNP (Experimental): Infusion of CNP prior to IR injury
  Interventions: Drug: C-type natriuretic peptide (CNP); Drug: Acetylcholine
- Saline (Placebo Comparator): Effect of saline infusion prior to IR injury
  Interventions: Drug: Saline; Drug: Acetylcholine

INTERVENTIONS:
Drug: C-type natriuretic peptide (CNP) — 360 pmol/min for 15 minutes intra-arterially
  Arms: CNP
Drug: Saline — Sodium Chloride 0.9% intra-arterially 0.5ml/min
  Arms: Saline
Drug: Acetylcholine — 2 stepped infusions for a total 9min per limb, totalling 1.05micromoles per limb

SUMMARY:
To determine the effects of whether increasing CNP concentrations slightly above normal will improve the functioning of blood vessels after the interruption in the flow of blood. In this study we are looking at the function of the blood vessels of the forearm, as a substitute for those in the heart

ELIGIBILITY:
Inclusion Criteria:

* Healthy human volunteers on no systemic medication, excepting the oral contraceptive pill

Exclusion Criteria:

* History of medical illness
* Unwillingness to sign consent form
* Use of non-OCP medications
* Hypertension on examination of the blood pressure

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in area under curve dose-response to acetylcholine after IR injury | 2h

CONTACTS AND LOCATIONS:
Overall Officials: Ahluwalia Amrita, BSc PhD, Principal Investigator — Queen Mary University London
Locations (1):
- Queen Mary University London, London, United Kingdom